CLINICAL TRIAL: NCT02813200
Title: Description of the Ability to Learn How to Handle Inhaler Devices in COPD
Acronym: INTUITIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2014/22
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, inhaler device, handling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Drug: Seretide® Diskus® 500/550 μg; Drug: Ultibro® Breezhaler® 110/50 μg; Drug: Spiriva® Respimat® 2,5 μg
- Group 2 (Experimental)
  Interventions: Drug: Seretide® Diskus® 500/550 μg; Drug: Ultibro® Breezhaler® 110/50 μg; Drug: Spiriva® Respimat® 2,5 μg
- Group 3 (Experimental)
  Interventions: Drug: Seretide® Diskus® 500/550 μg; Drug: Ultibro® Breezhaler® 110/50 μg; Drug: Spiriva® Respimat® 2,5 μg

INTERVENTIONS:
Drug: Seretide® Diskus® 500/550 μg — Every day during 7 days
Drug: Ultibro® Breezhaler® 110/50 μg — Every day during 7 days
Drug: Spiriva® Respimat® 2,5 μg — Every day during 7 days

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the fourth leading cause of death in the world and further increase in its prevalence and mortality has been predicted. Currently, the main long-term treatments are the long-acting beta-2 agonist, indacaterol, salmeterol and the anticholinergic drug, tiotropium and glycopyrronium, used alone or in combination:

* long-acting beta-2 agonist with corticosteroid (e.g. salmeterol/fluticasone),
* long-acting beta-2 agonist with anticholinergic (e.g. indacatetrol/glycopyrronium).

These drugs are delivered to the lung using different inhaler devices such as Breezhaler ®, Handihaler® and Diskus®.

DETAILED DESCRIPTION:
The correct use of inhaler devices is an inclusion criterion in COPD clinical trials. In real life, patients may make many errors using their own inhaler device, which may alter the positive effects observed in clinical trials.

The main objective of this study is to describe the handling of inhaler devices (indacaterol-glycopyrronium Breezhaler®, tiotropium Respimat® and salmeterol-fluticasone Diskus®) in patients with COPD.

All participants will receive each of the three treatments (Seretide® Diskus® 500/550 μg, Ultibro® Breezhaler® 110/50 μg and Spiriva® Respimat® 2,5 μg). Each treatment will be given daily for one week, followed by a 7-day washout period.

On day 1 of each treatment period, the patient will have clinical examination, lung function testing (FEV1) and 2 video recordings:

* Video recording #1: inhalation (one puff) without any instruction of use,
* Video recording #2: inhalation (one puff) after reading the patient information leaflet.

At the end of the visit, the patient will watch a standardized video demonstrating correct inhaler technique.

On day 7 of each treatment period, the patient will have clinical examination, lung function testing (FEV1) and 1 video recording of inhaler device use (one puff).

30 days after the last visit, the patient will have a phone contact to collect the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 40 years,
* Written informed consent,
* Diagnosis of COPD according to international guidelines (GOLD 2012),
* Social security or health insurance,
* Women of childbearing potential with a very effective contraception according to the Haute Autorité de Santé (HAS) recommendations.

Exclusion Criteria:

* Previous treatment with Breezhaler®, Diskus® or Respimat® or similar device,
* QT ≥ 450 ms,
* Contraindications to tiotropium: hypersensitivity to tiotropium,
* Contraindications to indacatérol: hypersensitivity to indacatérol,
* Contraindications to salmeterol: hypersensitivity to salmeterol,
* Contraindications to fluticasone: hypersensitivity to fluticasone,
* Contraindications to glycopyrronium: hypersensitivity to glycopyrronium,
* COPD exacerbation within 6 weeks before inclusion,
* Chronic psychiatric disease,
* Medical condition that may affect handling of inhaler devices,
* Subject deprived of his/her liberty,
* Protected adult,
* Subject in exclusion period related to another protocol,
* Pregnant or breastfeeding woman

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the presence of at least a major error in the use of the inhalation system, from standardized checklist | Day 7 of each treatment

SECONDARY OUTCOMES:
Number of non critical errors from standardized checklist | Day 7 of each treatment
Number of non device-dependant errors from standardized checklist | Day 7 of each treatment
Measure of the time necessary for drug administration | Up to day 7 of each treatment
  Time in second
Measure of Forced Expiratory Volume in 1 second (FEV1) | At baseline and at day 7
Collection of adverse events | Up to day 66

CONTACTS AND LOCATIONS:
Overall Officials: Hélène PEYROUZET, Dr, Study Chair — Service Hospitalo-Universitaire de Pharmacologie Médicale
Locations (1):
- CIC-P - Centre François Magendie - G3 - Hôpital Haut-Lévêque, Bordeaux, France